CLINICAL TRIAL: NCT02149160
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Escalating, Phase 2a Safety, Tolerability, and Pharmacodynamic Study of Two Doses of an Histone Deacetylase Inhibitor (FRM-0334) in Subjects With Prodromal to Moderate Frontotemporal Dementia With Granulin Mutation
Brief Title: Study to Assess the Safety, Tolerability, and Pharmacodynamic (PD) Effects of FRM-0334 in Subjects With Prodromal to Moderate Frontotemporal Dementia With Granulin Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: FORUM Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FRM-0334-002; 2014-001489-85 (EudraCT Number)
Record Dates: First submitted 2014-05-20; First posted 2014-05-29 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2015-05

CONDITIONS: Granulin Mutation
Keywords: Histone deacetylase inhibitor; Frontotemporal dementia; Granulin
MeSH Terms: conditions — Frontotemporal Dementia | interventions — FRM-0334

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- FRM-0334; Arm 1 (Experimental): low dose, Capsule, Once Daily, Day 1 through Day 28
  Interventions: Drug: FRM-0334
- FRM-0334; Arm 2 (Experimental): high dose, Capsule, Once Daily, Day 1 through Day 28
  Interventions: Drug: FRM-0334
- Placebo Comparator; Arm 3 (Placebo Comparator): Placebo, Capsule, Once Daily, Day 1 through Day 28
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FRM-0334
  Arms: FRM-0334; Arm 1; FRM-0334; Arm 2
Drug: Placebo
  Arms: Placebo Comparator; Arm 3

SUMMARY:
The purposes of this study are to investigate the safety, tolerability, and pharmacodynamics of FRM-0334 in subjects with prodromal to moderate frontotemporal dementia with granulin mutation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ages aged ≥21 and ≤75 years
* Genotyped positive for a FTD-GRN mutation, and aware of it
* Prodromal to moderate FTD-GRN
* Resides in a stable living situation, living at home, senior residential setting, or an institutional setting without the need for continuous (ie, 24-hour) nursing care
* Proficiency (oral and written) in the language in which study-related documents, including the ICF and standardized tests, will be administered
* Able to swallow capsules
* Be in good general health, willing and able to comply with the protocol requirements, and expected to complete the study as designed (in the judgment of the investigator)

Exclusion Criteria:

* Clinically significant abnormalities on physical examination, medical history, ECG, vital signs, laboratory values, or unstable medical or psychiatric illness
* Females who are pregnant, breastfeeding, or planning to become pregnant during the study

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of FRM-0334 | Baseline to Day 28 or Early Termination
  * Number and percentage of subjects with AEs
  * Number and percentage of subjects with SAEs
  * Number and percentage of subjects who discontinue due to AEs
  * Number and percentage of subject deaths
Assess the pharmacodynamic (PD) effects of FRM-0334 on the change from baseline in plasma concentrations of progranulin (PGRN) after 28 days | Baseline to Day 28 or Early Termination

SECONDARY OUTCOMES:
Assess the pharmacodynamic effects of FRM-0334 on the change from baseline in cerebrospinal fluid (CSF) concentrations of PGRN after 28 days | Baseline and Day 28
  Change in CSF progranulin concentration from baseline
Characterize the plasma concentrations of FRM-0334 and metabolites following once daily dosing for 28 days | Day 1 to Day 28 or Early Termination
  Cmax, Ctrough, tmax, t1/2, λz, AUC(0-τ), CL/F, Cav in plasma
Characterize the CSF concentrations of FRM-0334 and metabolites following once daily dosing for 28 days | Day 1 to Day 28 or Early Termination
  Cmax, Ctrough, tmax, t1/2, AUC0-τ, CL/F, Cav in CSF

CONTACTS AND LOCATIONS:
Locations (13):
- United States (5):
  - UCSF Memory and Aging Center, San Francisco, California
  - Compass Research, LLC, Orlando, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Perelman School of Medicine, University of Pennsylvania, Philadelphia, Pennsylvania
- University Hospitals Leuven, Leuven, Belgium
- France (2):
  - CHU Bordeaux Hospital Pellegrin, Bordeaux
  - CHU Rouen, Charles Nicolle Hospital, Rouen
- Italy (3):
  - IRCCS - Centro S. Giovanni di Dio FateBeneFratelli, Brescia
  - Neurological Clinic, University of Brescia, AO Civil Hospital of Brescia, Brescia
  - Fondazione Universita Gabriele D'Annunzio di Chieti, Chieti Scalo
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands
- The National Hospital for Neurology and Neuroscience, London, United Kingdom

REFERENCES:
- [Derived] Ljubenkov PA, Edwards L, Iaccarino L, La Joie R, Rojas JC, Koestler M, Harris B, Boeve BF, Borroni B, van Swieten JC, Grossman M, Pasquier F, Frisoni GB, Mummery CJ, Vandenberghe R, Le Ber I, Hannequin D, McGinnis SM, Auriacombe S, Onofrj M, Goodman IJ, Riordan HJ, Wisniewski G, Hesterman J, Marek K, Haynes BA, Patzke H, Koenig G, Hilt D, Moebius H, Boxer AL. Effect of the Histone Deacetylase Inhibitor FRM-0334 on Progranulin Levels in Patients With Progranulin Gene Haploinsufficiency: A Randomized Clinical Trial. JAMA Netw Open. 2021 Sep 1;4(9):e2125584. doi: 10.1001/jamanetworkopen.2021.25584. PMID 34559230